CLINICAL TRIAL: NCT00811265
Title: Safety, Compatibility and Imaging Quality of ExAblate Prostate Applicator for Prostate Cancer
Brief Title: Safety Evaluation of ExAblate MRgFUS for Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC001
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
Keywords: ExAblate MRgFUS; Focused ultrasound; Magnetic resonance imaging; Prostate cancer; Radical prostatectomy candidate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simulated ExAblate MRgFUS (Experimental): Patients undergoing simulated ExAblate MRgFUS device use
  Interventions: Device: ExAblate MRgFUS for prostate cancer

INTERVENTIONS:
Device: ExAblate MRgFUS for prostate cancer — Simulated use of ExAblate MRgFUS system

SUMMARY:
Evaluate the safety, compatibility and imaging quality of the ExAblate MRgFUS system.

DETAILED DESCRIPTION:
The objective of this study is to evaluate safety, compatibility and imaging quality of the ExAblate MRgFUS system for prostate cancer, under simulated use conditions. No acoustic energy will be delivered and no focused ultrasound therapy will be performed. This is an imaging only study.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients: up to 75 years.
* Men scheduled for radical prostatectomy due to prostate cancer.
* Patients who are able and willing to give consent and able to attend all study visits.

Exclusion Criteria:

* Contraindications to MRI including: claustrophobia, weight over 120 kg, implanted ferromagnetic materials or foreign objects, and known intolerance to the MRI contrast agent (e.g. Gadolinium or Magnevist)
* Severely abnormal coagulation (INR>1.5)
* Patients with unstable cardiac status including: unstable angina pectoris on medication, patients with documented myocardial infarction within six months of protocol entry, congestive heart failure requiring medication (other than diuretic), patients on anti-arrhythmic drugs, severe hypertension (diastolic BP > 100 on medication), and patients with cardiac pacemakers
* Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during imaging (approximately 1 hrs.)
* Any rectal pathology preventing probe insertion, (as active proctitis, ulcerative colitis, fissure ani, diverticulitis, previous rectal surgery, IBD, etc…)
* Any spinal pathology that prohibits maintaining supine position for more then an hour
* Any previous radiation to the pelvis.

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Device-related adverse events | Throughout study period

SECONDARY OUTCOMES:
Device compatibility with human anatomy | During simulated device use
MR Imaging Quality | During simulated device use

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- See also: Web page of clinical study Sponsor — http://www.insightec.com